CLINICAL TRIAL: NCT05425433
Title: Should Serial Casting be a "First-resort" Conservative Treatment for Adults With Upper Extremity Burn Contractures?
Brief Title: Serial Casting for Upper Extremity Burn Contractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22.084
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Burn Contracture of Skin
Keywords: Burns, Burn Rehabilitation, Serial Casting
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serial casted joint (Experimental): Tailored serial casting intervention following 1 week of usual care
  Interventions: Other: Tailored serial casting intercention

INTERVENTIONS:
Other: Tailored serial casting intercention — Every participant will undergo 1 week of usual care for the affected joint according to the OT's prescription (static progressive, dynamic or serial static) combined with stretching, moisturizers, pressure therapy, or thermal modalities. After the one week of splinting, if the PROM of the targeted joint does not improve, the participant will start serial casting (Monday to Friday). Patients will have a cast applied on Monday morning and worn for 24hrs/day or for 48hrs according to the OTs and treating physician's decision (rationale documented).The OT will decide how many weeks the participant will be wearing casts and the rationale to stop this treatment will be documented. When the treatment is stopped, patients will be encouraged to wear a maintenance splint for the following 2 weeks.

SUMMARY:
The use of a splint, serial casting and passive stretching have been described in the literature as conservative interventions to manage joint contractures after burn injury. There is a paucity of literature investigating the effect of serial casting on scar contractures following upper extremity (UE) burn injury in adults and a lack of studies using strong methodological approaches. There are also no studies investigating the effect of casting on hypertrophic scars (HSc) and on self-reported UE function. This study is a longitudinal case series design with a criteria for change on the use of serial casting for the treatment of upper extremity burn contractures. The purpose of this study is to estimate the extent to which range of motion (AROM and PROM), scar characteristics and patient-reported upper-extremity function changes following an individually-tailored serial casting treatment program after switching from one week of usual care and to determine if these changes can be maintained 3 weeks after stopping serial casting, for adult burn survivors who developed an upper-extremity joint contracture greater than 15% normal range of motion within 1-year post-burn. This study will be a longitudinal case series design with a criteria for change. A minimum of 12 participants will be recruited from the "Centre d'expertise pour les victimes de brûlures graves de l'ouest du Québec" (CEVBGOQ) and will undergo one week of "usual care". If the PROM of the joint does not improve after one week of usual care, the participant will start the serial casting process, which will be prescribed by the treating OT. PROM/AROM and scar characteristics will be measured using a revised goniometry protocol that incorporates cutaneokinematics (CKM) principles and precise skin measures (DermaScan C, Cutometer®, Mexameter® and Tewameter®) at baseline, every Monday and Friday of the treatment weeks and 3 weeks after treatment cessation. Self-reported UE function and satisfaction related to scarring will be assessed at baseline and 3 weeks after treatment cessation using the QuickDASH and the patient satisfaction assessment scale (PSAS). Analysis on ROM and scar characteristic will be conducted using a graphical representation with a projected "usual care" regression line to count how many outcomes were over the line once the treatment was introduced. This study will contribute to building evidence for the use of serial casting following UE burn contractures in the adult population.

DETAILED DESCRIPTION:
Participants will undergo a tailored intervention based on their needs.

ELIGIBILITY:
Inclusion Criteria:

* Burn survivors with >15% loss of PROM of their PIP, MCP, wrist, or elbow in either: flexion, extension, ulnar deviation or radial deviation.
* Fire, flame or scald burn injury

  -≥16 years old
* have provided informed consent.

Exclusion Criteria:

* Frostbite, chemical or electrical burn injury
* A premorbid musculoskeletal or neurological disorder that limited their ROM
* Have sustained a neurological injury secondary to the burn injury
* A psychiatric or cognitive disorder that limits their ability to follow the research protocol
* Have been diagnosed with heterotopic ossification
* PROM is contraindicated for any reason
* Do not understand English or French.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Passive range of motion changes | Baseline, Every Monday and Friday of Serial casting intervention weeks (tailored to the patient's needs), 3 weeks post intervention
  PROM measures by goniometer (standard and revised goniometry protocol)
Active range of motion changes | Baseline, Every Monday and Friday of Serial casting intervention weeks (tailored to the patient's needs), 3 weeks post intervention
  AROM measures by goniometer (standard and revised goniometry protocol)

SECONDARY OUTCOMES:
Patient reported upper-extremity function changes | Baseline, 3 weeks post intervention
  Short version of The Disabilities of the Arm, Shoulder and Hand questionnaire (QuickDASH); A higher score indicates a greater level of disability and severity, whereas, lower scores indicates a lower level of disability. The score ranges from 0 (no disability) to 100 (most severe disability).
Scar patient satisfaction | Baseline, 3 weeks post intervention
  Patient satisfaction assessment scale (PSAS), A higher score indicates a lower satisfaction towards the scar. The score ranges from 6 (Very satisfied) to60 (Not satisfied at all).
Skin Thickness Changes | Baseline, Every Monday and Friday of Serial casting intervention weeks (tailored to the patient's needs), 3 weeks post intervention
  Ultrasound skin measures, mm
Skin Elasticity Changes | Baseline, Every Monday and Friday of Serial casting intervention weeks (tailored to the patient's needs), 3 weeks post intervention
  Skin elasticity measures (r0- Cutometer), mm
Skin Erythema Changes | Baseline, Every Monday and Friday of Serial casting intervention weeks (tailored to the patient's needs), 3 weeks post intervention
  Erythema index measure by Mexameter, scale values of 0 to 999. The erythema values are individual for each person and depend strongly on the ethnic group. The measurements are generally used to determine changes before and after a treatment.
Skin Melanin Changes | Baseline, Every Monday and Friday of Serial casting intervention weeks (tailored to the patient's needs), 3 weeks post intervention
  Melanin index measured by Mexameter
Trans-epidermal water loss (TEWL) | Baseline, Every Monday and Friday of Serial casting intervention weeks (tailored to the patient's needs), 3 weeks post intervention
  Trans-epidermal water loss (TEWL) measured by Tewameter

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Nedelec, PhD, Principal Investigator — CRCHUM
Locations (1):
- Hôpital de réadaptation Villa Médica, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided